CLINICAL TRIAL: NCT02391337
Title: Evaluating Different Rate Control Therapies in Permanent Atrial Fibrillation: A Prospective, Randomised, Open-label, Blinded Endpoint Feasibility Pilot Comparing Digoxin and Beta-blockers as Initial Rate Control Therapy
Brief Title: Rate Control Therapy Evaluation in Permanent Atrial Fibrillation (RATE-AF)
Acronym: RATE-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBCCS_RATEAF
Record Dates: First submitted 2015-02-27; First posted 2015-03-18 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Permanent Atrial Fibrillation
Keywords: Atrial fibrillation; Quality of life; Left ventricular ejection fraction; Diastolic function; Echocardiography; Beta-blockers; Digoxin
MeSH Terms: conditions — Atrial Fibrillation | interventions — Bisoprolol; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-blocker (Active Comparator): In Group B, oral bisoprolol will be commenced at either 1.25mg, 2.5mg or 5mg according to the treatment schedule and uptitrated, as required, to 15mg daily. Recommended additional therapy in this arm includes diltiazem. Use of digoxin is explicitly discouraged but will not terminate participation in the study. If intolerance to bisoprolol occurs, investigators will be advised to try an alternate beta-blocker of their choosing (typically carvedilol, nebivolol, or metoprolol) at equivalent dosage.
  Interventions: Drug: Bisoprolol
- Digoxin (Active Comparator): In Group A, the maintenance dose of oral digoxin will be either 62.5mcg or 125mcg according to the pre-defined treatment schedule and uptitrated, as required, to 250mcg daily. A single loading dose of four tablets (250 or 500mcg according to target maintenance dose) will be prescribed in digoxin-naïve participants, where necessary. Recommended additional therapy in this arm includes the calcium-channel blocker diltiazem. Use of beta-blockers is explicitly discouraged but will not terminate participation in the study.
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Bisoprolol — Drug intervention
  Arms: Beta-blocker
Drug: Digoxin — Drug intervention
  Arms: Digoxin

SUMMARY:
Atrial fibrillation is a common heart rhythm disturbance, causing important discomfort for patients, a high risk of stroke, frequent hospital admissions and a two-fold increase in death. The number of patients with this condition are expected to double in the next 20 years. Medications to control heart-rate are used in the majority of patients, although the choice of agent is often guided by local preference rather than evidence from controlled trials. Despite the fact that patients with atrial fibrillation have high rates of other cardiac conditions such as heart failure, clinicians have insufficient evidence to personalise the use of different therapies. This feasibility study will allow us to develop a range of methods that can characterise patients according to the pumping and relaxing function of the heart, the burden of symptoms and to identify new blood markers. In this way, the investigators hope to improve clinical practice guidelines, allowing doctors to prescribe appropriate treatments for the right patients.

The research will be focused around a randomised trial of two medication strategies, providing much-needed data on the comparison of digoxin and beta-blockers (two commonly-used drugs in patients with atrial fibrillation). It will also allow us to identify the best way to record patient-reported quality of life and develop robust techniques to determine heart function using non-invasive imaging, facilitating the conduct of a large-scale clinical trial. The key objectives of the research programme are to define the optimal medications for patients with atrial fibrillation and identify the most valid, reproducible and cost-effective methods to examine patients. The ultimate aim of the project is to improve clinical outcomes in atrial fibrillation, benefiting patients, the National Health Service and the global community.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is an increasingly common cardiac condition that leads to a substantial burden on quality-of-life (QoL), an increased risk of cardiovascular events, hospitalisation and death, and significant healthcare costs for the NHS. In addition to anti-coagulation and considerations for rhythm control therapy, most patients with AF are in need of pharmacological control of heart rate. This aspect of care has not received stringent investigation, with treatment guidelines based on small crossover studies and observational data rather than robust controlled trials. Beta-blocker monotherapy remains the first-line option in the current NICE AF guidelines consultation document, with digoxin only for sedentary patients, although this recommendation is based on 'very low-quality evidence'. The benefit of different rate-control therapies on symptoms and other intermediate outcomes (such as left-ventricular ejection fraction [LVEF] and diastolic function) are unknown, as are their effects on clinical events such as hospitalisation. This situation is unacceptable in light of the potential benefits and risk of different rate-control options in AF. It also limits our ability to personalise treatment according to patient characteristics.

The RAte control Therapy Evaluation in permanent Atrial Fibrillation (RATE-AF) trial is informed by a number of in-depth systematic reviews of management and clinical outcomes in AF patients. Taken together, this information provides a sound basis to plan a major randomised controlled trial (RCT). However as trials of rate-control in AF have typically been small or uncontrolled, further information is needed before designing a trial that can assess clinical outcomes. The RATE-AF trial will allow us to define appropriate primary and secondary outcome measures and their standard deviation in a contemporary population of patients with permanent AF. This information will allow us to estimate sample size, determination of recruitment, retention and adherence policies, and to ascertain the best methods of obtaining adverse event data and reliable economic costs for a larger trial assessing cardiovascular outcomes and hospitalization. The RATE-AF trial will also be the largest RCT of its kind, allowing us to compare the effect of beta-blockers and digoxin on QoL as initial rate-control therapy in patients with permanent AF. The long-term aim of the research is to answer key questions about how to initiate therapy, stratified by relevant patient characteristics such as systolic and diastolic cardiac function, baseline symptoms and concurrent medication. The research will also define the patho-physiological mechanisms underlying AF-related symptoms, left-ventricular function and their association with adverse clinical outcomes, and to identify clinical markers for the response to different rate control therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 60 years or older, able to provide informed written consent
2. Permanent AF, characterised (at time of randomisation) as a physician decision for rate-control with no plans for cardioversion, anti-arrhythmic medication, or ablation therapy
3. Symptoms of breathlessness (New York Heart Association Class II or more)
4. Able to provide written, informed consent

Exclusion Criteria:

1. Established indication for beta-blocker therapy, e.g. survived myocardial infarction in the last 6 months
2. Known contraindications for therapy with beta-blockers or digoxin, e.g. a history of severe bronchospasm that would preclude use of beta-blockers, or known intolerance to these medications
3. Baseline heart rate <60 bpm
4. Known intolerance of beta-blockers or digoxin
5. A history of severe bronchospasm (e.g. due to asthma) that would preclude use of beta-blockers
6. Baseline heart rate <60 bpm
7. History of second or third-degree heart block
8. Supraventricular arrhythmias associated with accessory conducting pathways (e.g. Wolff-Parkinson-White syndrome) or a history of ventricular tachycardia or fibrillation
9. Planned pacemaker implantation, pacemaker-dependent rhythm or history of atrioventricular node ablation
10. Decompensated heart failure (evidenced by need for intravenous inotropes, vasodilators or diuretics) within 14 days prior to randomisation
11. A current diagnosis of hypertrophic cardiomyopathy, myocarditis or constrictive pericarditis
12. Received or on waiting list for heart transplantation
13. Initiation of cardiac resynchronization therapy (with/without defibrillator) within 6 months prior to randomisation
14. Intravenous infusions for heart failure (inotropes, vasodilators or diuretics) within 7 days prior to randomisation
15. A current diagnosis of hypertrophic cardiomyopathy, myocarditis or constrictive pericarditis
16. Received or on waiting list for heart transplantation
17. Receiving renal replacement therapy
18. Major surgery, including thoracic or cardiac surgery, within 3 months of randomisation
19. Severe, concomitant non-cardiovascular disease (including malignancy) that is expected to reduce life expectancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dipak Kotecha, MBChB PhD MRCP, Principal Investigator — University of Birmingham
Locations (2):
- United Kingdom (2):
  - City Hospital, Birmingham, West Midlands
  - Queen Elizabeth Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotecha D, Holmes J, Krum H, Altman DG, Manzano L, Cleland JG, Lip GY, Coats AJ, Andersson B, Kirchhof P, von Lueder TG, Wedel H, Rosano G, Shibata MC, Rigby A, Flather MD; Beta-Blockers in Heart Failure Collaborative Group. Efficacy of beta blockers in patients with heart failure plus atrial fibrillation: an individual-patient data meta-analysis. Lancet. 2014 Dec 20;384(9961):2235-43. doi: 10.1016/S0140-6736(14)61373-8. Epub 2014 Sep 2. PMID 25193873
- [Derived] Akoumianakis I, Gilligan LC, Bunting KV, Fobian D, Kirchhof P, Arlt W, Taylor AE, Pavlovic D, Kotecha D; Rate control Therapy Evaluation in permanent Atrial Fibrillation (RATE-AF) trial team. Quantification and impact of circulating cardiotonic steroids in the RATE-AF randomised trial of patients with atrial fibrillation and heart failure. BMC Med. 2025 Dec 29;23(1):694. doi: 10.1186/s12916-025-04476-2. PMID 41462450
- [Derived] Abdali Z, Bunting KV, Mehta S, Camm J, Rahimi K, Stanbury M, Haynes S, Kotecha D, Jowett S. Cost-effectiveness of digoxin versus beta blockers in permanent atrial fibrillation: the Rate Control Therapy Evaluation in Permanent Atrial Fibrillation (RATE-AF) randomised trial. Heart. 2025 Mar 26;111(8):362-369. doi: 10.1136/heartjnl-2024-324761. PMID 39819610
- [Derived] Gill SK, Barsky A, Guan X, Bunting KV, Karwath A, Tica O, Stanbury M, Haynes S, Folarin A, Dobson R, Kurps J, Asselbergs FW, Grobbee DE, Camm AJ, Eijkemans MJC, Gkoutos GV, Kotecha D; BigData@Heart Consortium; cardAIc group; RATE-AF trial team. Consumer wearable devices for evaluation of heart rate control using digoxin versus beta-blockers: the RATE-AF randomized trial. Nat Med. 2024 Jul;30(7):2030-2036. doi: 10.1038/s41591-024-03094-4. Epub 2024 Jul 15. PMID 39009776
- [Derived] Kotecha D, Bunting KV, Gill SK, Mehta S, Stanbury M, Jones JC, Haynes S, Calvert MJ, Deeks JJ, Steeds RP, Strauss VY, Rahimi K, Camm AJ, Griffith M, Lip GYH, Townend JN, Kirchhof P; Rate Control Therapy Evaluation in Permanent Atrial Fibrillation (RATE-AF) Team. Effect of Digoxin vs Bisoprolol for Heart Rate Control in Atrial Fibrillation on Patient-Reported Quality of Life: The RATE-AF Randomized Clinical Trial. JAMA. 2020 Dec 22;324(24):2497-2508. doi: 10.1001/jama.2020.23138. PMID 33351042
- [Derived] Kotecha D, Calvert M, Deeks JJ, Griffith M, Kirchhof P, Lip GY, Mehta S, Slinn G, Stanbury M, Steeds RP, Townend JN. A review of rate control in atrial fibrillation, and the rationale and protocol for the RATE-AF trial. BMJ Open. 2017 Jul 20;7(7):e015099. doi: 10.1136/bmjopen-2016-015099. PMID 28729311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial opened for recruitment in December 2016 and the first participant was randomised on the 20th December 2016 and the last participant was randomised on the 1st October 2018. A total of 161 participants were randomised into the trial with 1 centre recruiting patients into the trial.
Pre-assignment Details: A total of 390 were screened for the trial, of these screened 161 were randomised.
Period: Baseline
Arm/Group | Beta-blocker | Digoxin
Started | 80 | 81
Completed | 80 | 81
Not Completed | 0 | 0
Period: 6 Months Follow-up
Arm/Group | Beta-blocker | Digoxin
Started | 80 | 81
Completed | 74 | 76
Not Completed | 6 | 5
Not completed — Death | 5 | 4
Not completed — Withdrawal by Subject | 1 | 1
Period: 12 Months Follow-up
Arm/Group | Beta-blocker | Digoxin
Started | 74 | 76
Completed | 72 | 73
Not Completed | 2 | 3
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beta-blocker | Digoxin | Total
Number analyzed (Participants) | 80 | 81 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.8 (8.1) | 74.4 (8.4) | 75.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 36 | 74
  Male | 42 | 45 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self declared ethnicity: White - English / Welsh / Scottish / Northern Iris | 66 | 72 | 138
  Self declared ethnicity: White-Irish | 8 | 4 | 12
  Self declared ethnicity: Asian / Asian British - Indian | 2 | 3 | 5
  Self declared ethnicity: Asian / Asian British - Pakistani | 3 | 0 | 3
  Self declared ethnicity: Black / African / Caribbean / Black British- African | 1 | 0 | 1
  Self declared ethnicity: Black / African / Caribbean / Black British - Caribbean | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 80 | 81 | 161
Creatinine [Mean (Standard Deviation); unit: Micromol/l] | 91.4 (23.1) | 87.9 (25.1) | 89.6 (24.1)
On anticoagulant before randomisation [Count of Participants; unit: Participants]
  No | 17 | 9 | 26
  Yes | 63 | 72 | 135
EHRA class [Count of Participants; unit: Participants] — Minimisation variables Note: EHRA Class was categorised into (Class 1, 2a) and (Class 2b, 3, 4) for the minimisation algorithm.
  The European Heart Rhythm Association score of atrial fibrillation (or EHRA score) is a classification system for the extent of atrial fibrillation.
  EHRA I - 'No symptoms' EHRA II - 'Mild symptoms'; normal daily activity not affected EHRA III - 'Severe symptoms'; normal daily activity affected EHRA IV - 'Disabling symptoms'; normal daily activity discontinued
  Participants
    EHRA Class 1 | 0 | 0 | 0
    EHRA Class 2a | 3 | 3 | 6
    EHRA Class 2b | 40 | 35 | 75
    EHRA Class 3 | 27 | 38 | 65
    EHRA Class 4 | 10 | 5 | 15
NYHA class [Count of Participants; unit: Participants] — NYHA Classification - The Stages of Heart Failure:
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    Class I | 0 | 0 | 0
    Class II | 53 | 47 | 100
    Class III | 24 | 32 | 56
    Class IV | 3 | 2 | 5
Previous diagnosis of heart failure? [Count of Participants; unit: Participants]
  No | 56 | 46 | 102
  Yes | 24 | 35 | 59
Any signs of heart failure at baseline [Count of Participants; unit: Participants]
  No | 45 | 32 | 77
  Yes | 35 | 49 | 84
Type I diabetes [Count of Participants; unit: Participants]
  No | 80 | 81 | 161
  Yes | 0 | 0 | 0
Type II diabetes [Count of Participants; unit: Participants]
  No | 58 | 65 | 123
  Yes | 22 | 16 | 38
Unplanned admission for AF or HF in last 12 months [Count of Participants; unit: Participants]
  No | 65 | 65 | 130
  Yes | 15 | 16 | 31
Any previous cardioversions [Count of Participants; unit: Participants]
  No | 71 | 74 | 145
  Yes | 9 | 7 | 16
Previously undergone AF ablation [Count of Participants; unit: Participants]
  No | 79 | 79 | 158
  Yes | 1 | 2 | 3
Previous history of anti-arrhythmic drugs [Count of Participants; unit: Participants]
  No | 72 | 75 | 147
  Yes | 8 | 6 | 14
Baseline NTproBNP [Median (Inter-Quartile Range); unit: pg/mL] | 1040.5 [752.5 to 1480] | 1091 [710 to 1522] | 1057 [744 to 1522]
Radial artery heart rate [Mean (Standard Deviation); unit: bpm] | 86.9 (10.3) | 87.8 (12) | 87.4 (11.2)
Apex beat heart rate [Mean (Standard Deviation); unit: bpm] | 99 (16.8) | 98.3 (15.1) | 98.7 (15.9)
12-Lead ECG Heart Rate [Mean (Standard Deviation); unit: bpm] | 99.2 (19.2) | 100.3 (16.8) | 99.7 (18)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 137.1 (17.5) | 134.5 (14.9) | 135.8 (16.2)
Estimated ejection fraction [Mean (Standard Deviation); unit: Percentage of ejection fraction] | 57.6 (10.5) | 56.2 (8.8) | 56.9 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Quality of Life (SF-36)
Description: Patient-reported outcomes as assessed by the SF-36 questionnaire physical component score.
  The physical component score ranges from 0-100 where higher value indicates better outcome.
Time Frame: Primary outcome at 6 months timepoint.
Population: ITT Analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 74 | 76
score on a scale | 29.7 (11.4) | 31.9 (11.7)

2. Secondary Outcome: Left Ventricular Ejection Fraction
Description: The above parameters will be measured using echocardiography and diastolic indices
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 72 | 73
percentage of ejection fraction | 59.8 (7.3) | 59.7 (8.7)

3. Secondary Outcome: Diastolic Function- Measured by the E/e'.
Description: The above parameters will be measured using echocardiography and diastolic indices.
  E/e' - the ratio between early mitral inflow velocity and mitral annular early diastolic velocity.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Ratio of E/e'
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 72 | 73
Ratio of E/e' | 10.8 (5.5) | 10.8 (5.1)

4. Secondary Outcome: B-type Natriuretic Peptide (BNP) at 6 Months.
Description: B-type natriuretic peptide (BNP) at 6 months.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 74 | 76
ng/L | 1209 [837 to 1531] | 1057.5 [625.5 to 1531]

5. Secondary Outcome: Composite Functional Status Measures- 6 Minute Walking Distance at 12 Months.
Description: Composite functional status measures- 6 minute walking distance at 12 months.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: metres
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 69 | 71
metres | 329 [120 to 429] | 366 [233 to 435]

6. Secondary Outcome: Patient Reported Outcomes- (AFEQT) at 12 Months.
Description: As assessed using the AFEQT overall score at 12 months. The range for AFEQT overall score is from 0= complete disability to 100=no disability.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 72 | 73
score on a scale | 68.1 (16.1) | 75.6 (17.1)

7. Secondary Outcome: Patient Reported Outcomes (SF36) Version 2 at 12 Months.
Description: As assessed using the SF-36 version 2 global and specific scores at 12 months. All domains presented are between 0 to 100 scale where the higher score indicates better outcomes.
Time Frame: 12 months
Population: Some domains of the SFF36 version 2 were not possible to be computed due to missing data in the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 72 | 73
score on a scale
  Physical Component Summary: number analyzed (Participants) | 72 | 72
  Physical Component Summary | 29.4 (12.4) | 32.5 (13)
  Mental Component Summary: number analyzed (Participants) | 72 | 72
  Mental Component Summary | 51.3 (10.1) | 53.6 (8.9)
  Physical Function Domain Score | 27.5 (13) | 31.5 (14.1)
  Role Limitation Due to Physical Domain score | 32 (12.4) | 37 (12.6)
  Role Limitation Due to Emotional Problems Domain score | 40.7 (15.5) | 45.2 (12.9)
  Social Functioning Domain Score | 43.3 (11.6) | 45.6 (12.3)
  Mental Health Domain | 51.8 (9.5) | 51.3 (9.3)
  Energy/Vitality Domain Score | 42 (10) | 47.1 (9.9)
  Pain Score | 41.9 (12.5) | 40.5 (12.7)
  General Health Perception Domain Score: number analyzed (Participants) | 72 | 72
  General Health Perception Domain Score | 39.6 (10) | 42.8 (9.9)

8. Secondary Outcome: Patient Reported Outcomes (EQ-5D-5L)
Description: As assessed using the EQ-5D-5L summary index questionnaires at both 6 and 12 months.
  The range for summary index is from -0.594=worst score to 1=best score
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 78 | 77
units on a scale | 0.62 (0.29) | 0.66 (0.27)

9. Secondary Outcome: Ambulatory Heart-rate.
Description: 24 hour ambulatory heart-rate.
Time Frame: Within 12 months
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 78 | 76
bpm | 73.7 (10.9) | 78.9 (11.3)

10. Other Pre Specified Outcome: Cardiovascular Events
Description: Number of Participants with hospital admissions for cardiovascular events.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 80 | 81
Participants | 12 | 2

11. Other Pre Specified Outcome: Drug Discontinuation Rate
Description: the number and extent to which patients discontinue trial drugs
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 72 | 73
Participants
  Adherent | 65 | 70
  Non-Adherent | 3 | 3
  Missing | 4 | 0

12. Other Pre Specified Outcome: Drug Discontinuation Rate Within 12 Months.
Description: Number of participants requiring drug discontinuation due to adverse reactions.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 80 | 81
Participants | 9 | 2

13. Other Pre Specified Outcome: Hospital Admission Rate
Description: A composite of adverse clinical events
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 80 | 81
Participants | 19 | 11

14. Other Pre Specified Outcome: Retention of Participants
Description: Convenience, compliance and cross-over data
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 80 | 81
Participants
  Death: yes | 7 | 4
  Death: No | 73 | 77
  Lost to follow-up: yes | 0 | 2
  Lost to follow-up: No | 80 | 79
  Withdrawn consent: yes | 1 | 2
  Withdrawn consent: No | 79 | 79

15. Other Pre Specified Outcome: Preferred Outcome Measures for This Cohort of Patients
Description: Establish which are the best measures for these patients
Time Frame: 12 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Population-specific Standard Deviations to Enable Sample Size Calculation for a Future Trial Powered to Detect a Difference in Hospital Admissions.
Description: SF-36 physical function score at 6 and 12 months
Time Frame: 12 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Population-specific Standard Deviations to Enable Sample Size Calculation for a Future Trial Powered to Detect a Difference in Hospital Admissions.
Description: SF-36 overall score at 6 and 12 months
Time Frame: 12 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Population-specific Standard Deviations to Enable Sample Size Calculation for a Future Trial Powered to Detect a Difference in Hospital Admissions.
Description: AFEQT overall score at 6 and 12 months
Time Frame: 12 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Population-specific Standard Deviations to Enable Sample Size Calculation for a Future Trial Powered to Detect a Difference in Hospital Admissions.
Description: LVEF and E/e scores at 6 and 12 months
Time Frame: 12 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Number of Participants With Unplanned Hospital Admissions.
Description: Number of Participants with Unplanned Hospital Admissions.
Time Frame: During the 12 month follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-blocker | Digoxin
Number analyzed (Participants) | 80 | 81
Participants | 19 | 11

ADVERSE EVENTS:
Time Frame: During the 12 month follow-up period.
Description: Adverse events (AEs) were recorded in the medical records and CRFs. Most AE/ARs that occurred in the trial, whether they are serious or not, were 'expected' treatment-related toxicities due to the drugs used in this trial.
Arm/Group | Beta-blocker | Digoxin
All-Cause Mortality (participants affected / at risk) | 7/80 | 4/81
Serious Adverse Events (participants affected / at risk) | 21/80 | 13/81
Other Adverse Events (participants affected / at risk) | 51/80 | 20/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beta-blocker (N=80) | Digoxin (N=81)
Cardiac Arrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac General (Cardiac disorders) | 4 (5) | 1 (2)
Haemorrhage/Bleeding (Vascular disorders) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 3 (5) | 1 (1)
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Constitutional Symptoms (General disorders) | 1 (1) | 1 (1)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain (Nervous system disorders) | 0 (0) | 1 (1)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Hepatobiliary/Pancreas (Hepatobiliary disorders) | 0 (0) | 1 (1)
Neurology (Nervous system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 4 (4) | 0 (0)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Renal/Genitourinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Vascular (Vascular disorders) | 2 (2) | 0 (0)
Lymphatics (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Death (Cardiac disorders) | 2 (2) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Death (Hepatobiliary disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Death (Renal and urinary disorders) | 1 (1) | 0 (0)
Death (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beta-blocker (N=80) | Digoxin (N=81)
Gastrointestinal upset (Gastrointestinal disorders) | 8 (8) | 5 (5)
Blurred vision (Eye disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Peripheral oedema (General disorders) | 11 (12) | 1 (1)
Symptomatic bradycardia (Cardiac disorders) | 5 (5) | 0 (0)
Dizziness (General disorders) | 24 (28) | 4 (4)
Headache (General disorders) | 9 (11) | 5 (5)
Lethargy (General disorders) | 30 (37) | 7 (7)
Upper respiratory tract symptoms (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 1 (1)
Symptomatic hypotension (Cardiac disorders) | 6 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT02391337/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02391337/SAP_001.pdf